CLINICAL TRIAL: NCT01588041
Title: Intraoperative OCT Guidance of Intraocular Surgery
Acronym: MIOCT
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00016827; R01EY023039 (NIH)
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Eye Manifestations
Keywords: Microscope mounted SDOCT
MeSH Terms: conditions — Eye Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (8):
- Vitreoretinal Interface Disease Group: A minimum of 50 subjects with vitreoretinal interface disease will be imaged with MIOCT prior to surgery, during surgical maneuvers, during a normal pause in surgery, and at 2 post-operative follow-up visits.
- Macular Hole Group: A minimum of 50 subjects with macular hole with be imaged with MIOCT prior to surgery, during surgical maneuvers, during a normal pause in surgery, and at 2 post-operative follow-up visits.
- Retinal Detachment Group: A minimum of 50 subjects with retinal detachment will be imaged with MIOCT prior to surgery, during surgical maneuvers, during a normal pause in surgery, and at 2 post-operative follow-up visits.
- Diabetic Retinopathy Group: A minimum of 50 subjects with diabetic retinopathy will be imaged with MIOCT prior to surgery, during surgical maneuvers, during a normal pause in surgery, and at 2 post-operative follow-up visits.
- Rare Related Macular Disease Group: Up to 70 subjects with rare related macular diseases will be imaged with MIOCT prior to surgery, during surgical maneuvers, during a normal pause in surgery, and at 2 post-operative follow-up visits.
- Generation 2 MIOCT Transition Group: 80 of the subjects recruited in years 1 through 5 (40 normal, 40 diseased) will be imaged with both the generation 1 MIOCT and the generation 2 MIOCT systems prior to surgery, during surgical maneuvers, during a normal pause in surgery, and at 2 post-operative follow-up visits.
- Endothelial Keratoplasty Group: 150 subjects undergoing Descemet Stripping Endothelial Keratoplasty (DSEK) will be imaged with MIOCT at the conclusion of the surgical procedure and may be imaged during follow-up visits.
- Anterior Lamellar Keratoplasty Group: 150 subjects undergoing Deep Anterior Lamellar Keratoplasty (DALK) will be imaged with MIOCT at the conclusion of the surgical procedure and may be imaged during follow-up visits.

SUMMARY:
The purpose of this study is to investigate the use of optical coherence tomography imaging integrated with an operating microscope (MIOCT) in ophthalmic surgeries.

DETAILED DESCRIPTION:
Optical Coherence Tomography (OCT) is used to capture reproducible ocular morphology and cross-sectional tissue measurements in-vivo in a rapid, non-invasive, non-contact manner. It has displaced ophthalmoscopy and stereo photography for clinical assessment and documentation of retinal microanatomy including thickness, cystoid structures, subretinal fluid and retinal traction.(1) Spectral Domain Optical Coherence Tomography (SDOCT) has the speed and resolution required for real-time noninvasive three-dimensional imaging of critical pathology.

While modern ophthalmic surgery has benefited from rapid advances in instrumentation and techniques (2-6), the basic principles of the stereo zoom operating microscope have not changed (except for increased automation) since the 1930's. (7-9) The ability to better resolve tissue microanatomy through real-time micro-imaging would have a dramatic impact on ophthalmic surgeon's capabilities, foster the development of new surgical techniques, and potentially improve surgical outcomes.

Complementary to microscope integrated OCT (MIOCT) testing, we use a commercial hand-held SDOCT instrument (Bioptigen, Inc.) during pauses in both anterior segment and retinal surgery to document surgical process.

While both the handheld instrument and Duke's Generation 1 (G1) MIOCT prototype have demonstrated that high-quality OCT imaging is possible during surgery, in both cases control of the OCT scan location and display of the real-time image data are managed on the OCT system console, located up to several feet from the surgeon. Thus, the potential dramatic impact of this technology on ophthalmic surgery is constrained by its limited integration with the surgical environment. The primary technical goal of this project is to address this issue through novel advances in OCT technology, automated tracking of surgical instruments and tools, and fusion of OCT controls, images and measurements into a seamless interface for the surgeon.

This study will facilitate future quality improvement processes based on intraoperative data matched to postoperative outcomes. Intraoperative OCT feedback will revolutionize communication in surgical research, clinical communication, surgeon training and continuing education, and will provide measurable data regarding disease patterns and intraoperative response, novel instrument and adjuvant use.

This study will prospectively examine the surgical utility of MIOCT in retinal and anterior segment surgery. A total of 722 subjects will be enrolled at 2 sites, Duke Eye Center and Cole Eye Institute. Of those, there will be 500 retina subjects and 222 anterior segment subjects. There will be a small number of normal subjects, who are not undergoing eye surgery, enrolled in this portion of this study for non-surgical study of the MIOCT system imaging, particularly for Generation 2 (G2) MIOCT. Rate of recruitment: 460 retina subjects will be enrolled at the rate of approximately 115 per year (~57 per year at both Duke and Cole) for years 1-4 and approximately 40 subjects will be enrolled in year 5 (adding up to a total of 500 subjects).

ELIGIBILITY:
Inclusion criteria

1. subjects undergoing surgery for vitreoretinal interface disease
2. subjects undergoing surgery for macular hole
3. subjects undergoing surgery for retinal detachment
4. subjects undergoing surgery for diabetic retinopathy with macular edema and/or traction detachments
5. subjects undergoing surgery for epiretinal membranes
6. subjects undergoing surgery for rare related macular diseases like myopic schisis.
7. subjects undergoing endothelial keratoplasty or anterior lamellar keratoplasty
8. subjects with normal ocular pathology enrolled as controls

Exclusion criteria:

1. Any ocular disease that restricts the ability to perform MIOCT scanning.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 722 subjects identified and recruited from the clinics of Duke Eye Center and Cole Eye Institute. Of those, there will be 500 retina subjects and 222 anterior segment subjects. Control subjects may include employees and students of both institutions.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2009-09; Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Test and provide feedback on the intraoperative system both in laboratory and then in the operating room. | 8.5 years
  The primary outcome of this project is to integrate optical coherence tomography (OCT) with the surgical environment through novel advances in OCT technology, automated tracking of surgical instruments and tools, and fusion of OCT controls, images and measurements into a seamless interface for the surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Toth, MD, Principal Investigator — Duke University Health System, Department of Ophthalmology; Joseph A Izatt, PhD, Principal Investigator — Duke University Department of Biomedical Engineering
Locations (2):
- United States (2):
  - Duke University Eye Center, Durham, North Carolina
  - Cole Eye Institute at the Cleveland Clinic Lemer College of Medicine, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All findings resulting from the MIOCT study will be prepared for publication in peer-reviewed journals and posted on PubMed Central once accepted. We are also strong advocates of open-access publishing whenever possible; one of the MPIs (Prof. Izatt) is the founding editor-in-chief of the Optical Society of America's (OSA) newest on-line, open-access journal Biomedical Optics Express (http://www.opticsinfobase.org/boe/home.cfm). We are supportive of efforts by publishers and professional societies to develop technologies for on-line publishing of entire experimental datasets. We have published such datasets using OSA's Interactive Science Publishing technology in the recent past (http://midas.osa.org/midaspub/item/view/1123).
  We will archive experimental results and findings from the proposed project for at least the duration of the project, and make the underlying datasets available to other researchers upon request.

REFERENCES:
- [Background] Mirza RG, Johnson MW, Jampol LM. Optical coherence tomography use in evaluation of the vitreoretinal interface: a review. Surv Ophthalmol. 2007 Jul-Aug;52(4):397-421. doi: 10.1016/j.survophthal.2007.04.007. PMID 17574065
- [Background] Machemer R. The development of pars plana vitrectomy: a personal account. Graefes Arch Clin Exp Ophthalmol. 1995 Aug;233(8):453-68. doi: 10.1007/BF00183425. No abstract available. PMID 8537019
- [Background] Tan DT, Mehta JS. Future directions in lamellar corneal transplantation. Cornea. 2007 Oct;26(9 Suppl 1):S21-8. doi: 10.1097/ICO.0b013e31812f685c. PMID 17881911
- [Background] Singh MS, MacLaren RE. Stem cells as a therapeutic tool for the blind: biology and future prospects. Proc Biol Sci. 2011 Oct 22;278(1721):3009-16. doi: 10.1098/rspb.2011.1028. Epub 2011 Aug 3. PMID 21813553
- [Background] Weiland JD, Cho AK, Humayun MS. Retinal prostheses: current clinical results and future needs. Ophthalmology. 2011 Nov;118(11):2227-37. doi: 10.1016/j.ophtha.2011.08.042. PMID 22047893
- [Background] Shin JY, Yu HG. Visual prognosis and spectral-domain optical coherence tomography findings of myopic foveoschisis surgery using 25-gauge transconjunctival sutureless vitrectomy. Retina. 2012 Mar;32(3):486-92. doi: 10.1097/IAE.0b013e31822058d1. PMID 21955988
- [Background] Machemer R, Parel JM. An improved microsurgical ceiling-mounted unit and automated television. Am J Ophthalmol. 1978 Feb;85(2):205-9. doi: 10.1016/s0002-9394(14)75949-5. PMID 623191
- [Background] Parel JM, Machemer R, Aumayr W. A new concept for vitreous surgery. 5. An automated operating microscope. Am J Ophthalmol. 1974 Feb;77(2):161-8. doi: 10.1016/0002-9394(74)90668-0. No abstract available. PMID 4812085
- [Background] Hahn P, Carrasco-Zevallos O, Cunefare D, Migacz J, Farsiu S, Izatt JA, Toth CA. Intrasurgical Human Retinal Imaging With Manual Instrument Tracking Using a Microscope-Integrated Spectral-Domain Optical Coherence Tomography Device. Transl Vis Sci Technol. 2015 Jul 1;4(4):1. doi: 10.1167/tvst.4.4.1. eCollection 2015 Jul. PMID 26175961
- [Background] Nam DH, Desouza PJ, Hahn P, Tai V, Sevilla MB, Tran-Viet D, Cunefare D, Farsiu S, Izatt JA, Toth CA. INTRAOPERATIVE SPECTRAL DOMAIN OPTICAL COHERENCE TOMOGRAPHY IMAGING AFTER INTERNAL LIMITING MEMBRANE PEELING IN IDIOPATHIC EPIRETINAL MEMBRANE WITH CONNECTING STRANDS. Retina. 2015 Aug;35(8):1622-30. doi: 10.1097/IAE.0000000000000534. PMID 25829349
- [Background] Kuo AN, Carrasco-Zevallos O, Toth CA, Izatt JA. Caveats to obtaining retinal topography with optical coherence tomography. Invest Ophthalmol Vis Sci. 2014 Sep 11;55(9):5730-1. doi: 10.1167/iovs.14-15212. No abstract available. PMID 25213121
- [Background] Folgar FA, Yuan EL, Farsiu S, Toth CA. Lateral and axial measurement differences between spectral-domain optical coherence tomography systems. J Biomed Opt. 2014 Jan;19(1):16014. doi: 10.1117/1.JBO.19.1.016014. PMID 24441877
- [Background] Kuo AN, McNabb RP, Chiu SJ, El-Dairi MA, Farsiu S, Toth CA, Izatt JA. Correction of ocular shape in retinal optical coherence tomography and effect on current clinical measures. Am J Ophthalmol. 2013 Aug;156(2):304-11. doi: 10.1016/j.ajo.2013.03.012. Epub 2013 May 6. PMID 23659972
- [Background] Hahn P, Migacz J, O'Donnell R, Day S, Lee A, Lin P, Vann R, Kuo A, Fekrat S, Mruthyunjaya P, Postel EA, Izatt JA, Toth CA. Preclinical evaluation and intraoperative human retinal imaging with a high-resolution microscope-integrated spectral domain optical coherence tomography device. Retina. 2013 Jul-Aug;33(7):1328-37. doi: 10.1097/IAE.0b013e3182831293. PMID 23538579
- [Background] Ehlers JP, Tao YK, Farsiu S, Maldonado R, Izatt JA, Toth CA. Visualization of real-time intraoperative maneuvers with a microscope-mounted spectral domain optical coherence tomography system. Retina. 2013 Jan;33(1):232-6. doi: 10.1097/IAE.0b013e31826e86f5. No abstract available. PMID 23190928
- [Background] Hahn P, Migacz J, O'Connell R, Izatt JA, Toth CA. Unprocessed real-time imaging of vitreoretinal surgical maneuvers using a microscope-integrated spectral-domain optical coherence tomography system. Graefes Arch Clin Exp Ophthalmol. 2013 Jan;251(1):213-20. doi: 10.1007/s00417-012-2052-2. Epub 2012 May 16. PMID 22585009
- [Background] Tao YK, Ehlers JP, Toth CA, Izatt JA. Intraoperative spectral domain optical coherence tomography for vitreoretinal surgery. Opt Lett. 2010 Oct 15;35(20):3315-7. doi: 10.1364/OL.35.003315. PMID 20967051
- [Background] Ehlers JP, Gupta PK, Farsiu S, Maldonado R, Kim T, Toth CA, Mruthyunjaya P. Evaluation of contrast agents for enhanced visualization in optical coherence tomography. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6614-9. doi: 10.1167/iovs.10-6195. Epub 2010 Nov 4. PMID 21051711
- [Background] Ehlers JP, Tao YK, Farsiu S, Maldonado R, Izatt JA, Toth CA. Integration of a spectral domain optical coherence tomography system into a surgical microscope for intraoperative imaging. Invest Ophthalmol Vis Sci. 2011 May 16;52(6):3153-9. doi: 10.1167/iovs.10-6720. PMID 21282565
- [Background] Hahn P, Migacz J, O'Connell R, Maldonado RS, Izatt JA, Toth CA. The use of optical coherence tomography in intraoperative ophthalmic imaging. Ophthalmic Surg Lasers Imaging. 2011 Jul;42 Suppl(0):S85-94. doi: 10.3928/15428877-20110627-08. PMID 21790116
- [Background] Ehlers JP, Kernstine K, Farsiu S, Sarin N, Maldonado R, Toth CA. Analysis of pars plana vitrectomy for optic pit-related maculopathy with intraoperative optical coherence tomography: a possible connection with the vitreous cavity. Arch Ophthalmol. 2011 Nov;129(11):1483-6. doi: 10.1001/archophthalmol.2011.316. PMID 22084218
- [Background] Pasricha ND, Shieh C, Carrasco-Zevallos OM, Keller B, Izatt JA, Toth CA, Kuo AN. Real-Time Microscope-Integrated OCT to Improve Visualization in DSAEK for Advanced Bullous Keratopathy. Cornea. 2015 Dec;34(12):1606-10. doi: 10.1097/ICO.0000000000000661. PMID 26509766
- [Background] Viehland C, Keller B, Carrasco-Zevallos OM, Nankivil D, Shen L, Mangalesh S, Viet du T, Kuo AN, Toth CA, Izatt JA. Enhanced volumetric visualization for real time 4D intraoperative ophthalmic swept-source OCT. Biomed Opt Express. 2016 Apr 12;7(5):1815-29. doi: 10.1364/BOE.7.001815. eCollection 2016 May 1. PMID 27231623
- [Background] Shen L, Carrasco-Zevallos O, Keller B, Viehland C, Waterman G, Hahn PS, Kuo AN, Toth CA, Izatt JA. Novel microscope-integrated stereoscopic heads-up display for intrasurgical optical coherence tomography. Biomed Opt Express. 2016 Apr 6;7(5):1711-26. doi: 10.1364/BOE.7.001711. eCollection 2016 May 1. PMID 27231616
- [Background] Seider MI, Tran-Viet D, Toth CA. MACULAR PSEUDO-HOLE IN SHAKEN BABY SYNDROME: UNDERSCORING THE UTILITY OF OPTICAL COHERENCE TOMOGRAPHY UNDER ANESTHESIA. Retin Cases Brief Rep. 2016 Summer;10(3):283-5. doi: 10.1097/ICB.0000000000000251. PMID 26655385
- [Background] Carrasco-Zevallos OM, Keller B, Viehland C, Shen L, Seider MI, Izatt JA, Toth CA. Optical Coherence Tomography for Retinal Surgery: Perioperative Analysis to Real-Time Four-Dimensional Image-Guided Surgery. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT37-50. doi: 10.1167/iovs.16-19277. PMID 27409495
- [Background] Todorich B, Shieh C, DeSouza PJ, Carrasco-Zevallos OM, Cunefare DL, Stinnett SS, Izatt JA, Farsiu S, Mruthyunjaya P, Kuo AN, Toth CA. Impact of Microscope-Integrated OCT on Ophthalmology Resident Performance of Anterior Segment Surgical Maneuvers in Model Eyes. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT146-53. doi: 10.1167/iovs.15-18818. PMID 27409466
- [Background] Grewal DS, Carrasco-Zevallos OM, Gunther R, Izatt JA, Toth CA, Hahn P. Intra-operative microscope-integrated swept-source optical coherence tomography guided placement of Argus II retinal prosthesis. Acta Ophthalmol. 2017 Aug;95(5):e431-e432. doi: 10.1111/aos.13123. Epub 2016 Jun 20. No abstract available. PMID 27321093
- [Background] Carrasco-Zevallos OM, Keller B, Viehland C, Shen L, Waterman G, Todorich B, Shieh C, Hahn P, Farsiu S, Kuo AN, Toth CA, Izatt JA. Live volumetric (4D) visualization and guidance of in vivo human ophthalmic surgery with intraoperative optical coherence tomography. Sci Rep. 2016 Aug 19;6:31689. doi: 10.1038/srep31689. PMID 27538478
- [Background] Grewal DS, Bhullar PK, Pasricha ND, Carrasco-Zevallos OM, Viehland C, Keller B, Shen L, Izatt JA, Kuo AN, Toth CA, Mruthyunjaya P. Intraoperative 4-Dimensional Microscope-Integrated Optical Coherence Tomography-Guided 27-Gauge Transvitreal Choroidal Biopsy for Choroidal Melanoma. Retina. 2017 Apr;37(4):796-799. doi: 10.1097/IAE.0000000000001326. PMID 27673716
- [Background] Pasricha ND, Shieh C, Carrasco-Zevallos OM, Keller B, Cunefare D, Mehta JS, Farsiu S, Izatt JA, Toth CA, Kuo AN. Needle Depth and Big-Bubble Success in Deep Anterior Lamellar Keratoplasty: An Ex Vivo Microscope-Integrated OCT Study. Cornea. 2016 Nov;35(11):1471-1477. doi: 10.1097/ICO.0000000000000948. PMID 27442318
- [Background] Pasricha ND, Bhullar PK, Shieh C, Carrasco-Zevallos OM, Keller B, Izatt JA, Toth CA, Freedman SF, Kuo AN. Four-dimensional Microscope-Integrated Optical Coherence Tomography to Visualize Suture Depth in Strabismus Surgery. J Pediatr Ophthalmol Strabismus. 2017 Feb 14;54:e1-e5. doi: 10.3928/01913913-20170201-01. PMID 28196266
- [Background] Chen X, Viehland C, Carrasco-Zevallos OM, Keller B, Vajzovic L, Izatt JA, Toth CA. Microscope-Integrated Optical Coherence Tomography Angiography in the Operating Room in Young Children With Retinal Vascular Disease. JAMA Ophthalmol. 2017 May 1;135(5):483-486. doi: 10.1001/jamaophthalmol.2017.0422. PMID 28384676
- [Background] Carrasco-Zevallos OM, Viehland C, Keller B, Draelos M, Kuo AN, Toth CA, Izatt JA. Review of intraoperative optical coherence tomography: technology and applications [Invited]. Biomed Opt Express. 2017 Feb 21;8(3):1607-1637. doi: 10.1364/BOE.8.001607. eCollection 2017 Mar 1. PMID 28663853
- [Background] Bhullar PK, Carrasco-Zevallos OM, Dandridge A, Pasricha ND, Keller B, Shen L, Izatt JA, Toth CA, Kuo AN. Intraocular Pressure and Big Bubble Diameter in Deep Anterior Lamellar Keratoplasty: An Ex-Vivo Microscope-Integrated OCT With Heads-Up Display Study. Asia Pac J Ophthalmol (Phila). 2017 Sep-Oct;6(5):412-417. doi: 10.22608/APO.2017265. PMID 28930381
- [Background] Qian R, Carrasco-Zevallos OM, Mangalesh S, Sarin N, Vajzovic L, Farsiu S, Izatt JA, Toth CA. Characterization of Long Working Distance Optical Coherence Tomography for Imaging of Pediatric Retinal Pathology. Transl Vis Sci Technol. 2017 Oct 16;6(5):12. doi: 10.1167/tvst.6.5.12. eCollection 2017 Oct. PMID 29057163
- [Background] Gabr H, Chen X, Zevallos-Carrasco OM, Viehland C, Dandrige A, Sarin N, Mahmoud TH, Vajzovic L, Izatt JA, Toth CA. VISUALIZATION FROM INTRAOPERATIVE SWEPT-SOURCE MICROSCOPE-INTEGRATED OPTICAL COHERENCE TOMOGRAPHY IN VITRECTOMY FOR COMPLICATIONS OF PROLIFERATIVE DIABETIC RETINOPATHY. Retina. 2018 Sep;38 Suppl 1(Suppl 1):S110-S120. doi: 10.1097/IAE.0000000000002021. PMID 29324591
- [Background] Hsu ST, Gabr H, Viehland C, Sleiman K, Ngo HT, Carrasco-Zevallos OM, Vajzovic L, McNabb RP, Stinnett SS, Izatt JA, Kuo AN, Toth CA. Volumetric Measurement of Subretinal Blebs Using Microscope-Integrated Optical Coherence Tomography. Transl Vis Sci Technol. 2018 Apr 5;7(2):19. doi: 10.1167/tvst.7.2.19. eCollection 2018 Apr. PMID 29651361
- [Background] Bleicher ID, Jackson-Atogi M, Viehland C, Gabr H, Izatt JA, Toth CA. Depth-Based, Motion-Stabilized Colorization of Microscope-Integrated Optical Coherence Tomography Volumes for Microscope-Independent Microsurgery. Transl Vis Sci Technol. 2018 Nov 1;7(6):1. doi: 10.1167/tvst.7.6.1. eCollection 2018 Nov. PMID 30405965